CLINICAL TRIAL: NCT01825590
Title: Effects of Simple Sodium Alignment on Short-, Medium- and Long-term Clinical and Laboratory Outcome Measures
Brief Title: Effects of Simple Sodium Alignment on Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 053-11
Record Dates: First submitted 2013-03-13; First posted 2013-04-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Complication of Hemodialysis
Keywords: hemodialysis; dialysate and serum sodium
MeSH Terms: interventions — Dialysis Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects undergoing sodium alignment: Dialysate and serum sodium concentration aligned
  Interventions: Other: Dialysate and serum sodium concentration aligned
- Subjects not undergoing sodium alignment: Dialysate and serum sodium concentration not aligned

INTERVENTIONS:
Other: Dialysate and serum sodium concentration aligned
  Groups: Subjects undergoing sodium alignment

SUMMARY:
A difference between dialysate and serum sodium concentration leads to diffusive sodium transfer across the dialyzer membrane. The consequences of diffusive sodium flux into the patient can be chronic sodium overload leading to overhydration, hypertension, cardiovascular disease, and other problems. Diffusive sodium flux out of the patient can lead to intradialytic blood pressure instability. A simple strategy for alignment of dialysate and serum sodium concentrations was implemented starting in April/May 2010 in order to minimize the problems particularly associated with chronic sodium overload.

DETAILED DESCRIPTION:
The purpose of this database analysis is to assess the impact that this operational change has had in the short, medium and long term on key clinical and laboratory parameters in the patients, including blood pressure, body weight, interdialytic weight gain, serum electrolytes, intradialytic saline administration, missed treatments, hospitalizations, medication, inflammatory markers, etc. All subjects included in the final dataset will be matched with dialysis patients receiving treatment in other dialysis clinics of the Renal Research Institute who were not subject to the operational change. This will lead to the development of a matched cohort of equal size unexposed to dialysate to serum sodium alignment.

The analysis is planned to investigate treatment effects, and test the effects of dialysate to serum sodium alignment for interactions and associations between those laboratory and clinical parameters. The extent and magnitude of sodium alignment (the operational change) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on hemodialysis

Exclusion Criteria:

* None

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects on hemodialysis
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Interdialytic weight gain | Each dialysis treatment (3x per week) - 2 years of treatment data
Pre-dialysis Blood Pressure | Each dialysis treatment (3x per week)- 2 years of treatment data

SECONDARY OUTCOMES:
Hospitalization rate and number of days | Per occurence during the entire follow-up period of 2 years

OTHER OUTCOMES:
Body weight | Each treatment (3x per week)- 2 years of treatment data
Serum electrolytes | Each treatment (3x per week)- 2 years of treatment data
Intradialytic saline administration | Per occurance
Inflammatory markers | Each treatment (3x per week)- 2 years of treatment data
Medications | Per occurance
Missed treatments | Per occurance

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States

REFERENCES:
- [Derived] Raimann JG, Ficociello LH, Usvyat LA, Zhang H, Pacelli L, Moore S, Sheppard P, Xiao Q, Wang Y, Mullon C, Balter P, Sullivan T, Kotanko P. Effects of dialysate to serum sodium (Na+) alignment in chronic hemodialysis (HD) patients: retrospective cohort study from a quality improvement project. BMC Nephrol. 2018 Apr 2;19(1):75. doi: 10.1186/s12882-018-0870-0. PMID 29609536